CLINICAL TRIAL: NCT05416515
Title: Phase 2 Clinical Trial of FIsetin to Treat CArpal Tunnel Syndrome (FITCATS)
Brief Title: A Study of Fisetin to Treat Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter C. Amadio, M.D. (Other)
Responsible Party: Sponsor-Investigator, Peter C. Amadio, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-010406
Record Dates: First submitted 2022-05-22; First posted 2022-06-13 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — fisetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carpal Tunnel Syndrome (Experimental): Adult men and women who have a clinical diagnosis for Carpal Tunnel Syndrome (CTS) will receive Fisetin for 2 day periods for 2 months
  Interventions: Drug: Fisetin

INTERVENTIONS:
Drug: Fisetin — 100 mg capsules orally for 2 consecutive days and, after 1 month, another 2 consecutive days

SUMMARY:
This research study is being conducted to investigate the safety and effectiveness of the drug Fisetin for mild or moderate carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
FITCATS trial will enroll approximately 40 subjects with mild-moderate CTS and evidence of senescence from blood markers into a short term (180 days) prospective phase 2 study of Fisetin therapy, using as outcome measures a well-accepted patient reported outcome questionnaire (Boston CTS questionnaire, BCTQ) as well as reduction from baseline in senescence markers in the blood, including SASP factors and inflammatory markers. Based on the known performance of the BCTQ, the investigators estimate that a sample size of 40 will be sufficient to show a clinically important difference in outcome, if it is present. Each subject will be enrolled for a six-month period. Subjects may withdraw at any time, for any reason.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria to be eligible for enrollment:

Inclusion Criteria:

* Males and females between age 21 and 80 years of age.
* Symptoms of numbness or tingling for at least 4 weeks in at least two digits on one hand that include thumb, index, long, or radial border of ring finger.
* Classic or probable carpal tunnel syndrome on Katz-Stirrat hand diagram.
* A clinical diagnosis of carpal tunnel syndrome. Patients with bilateral CTS will have the more severe hand enrolled.
* Able to complete English-language questionnaires and clinical evaluations.
* Willingness to avoid pregnancy.

  * Female participants of childbearing potential must have a negative pregnancy test at screening (serum) and before the first dose on Day 1 (urine), before the third dose on Day 29 (urine), and 60 days after the final dose on day 60 (urine).
  * Sexually active female participants of childbearing potential must agree to take appropriate precautions to avoid pregnancy from screening until 30 days after the last dose of study drug (day 60). Permitted methods in preventing pregnancy (see Appendix A) will be communicated to the participants and their compliance confirmed.
  * All female participants of childbearing potential will refrain from donating oocytes from screening-day 60 of the study.
  * Women without child bearing potential (ie., surgically sterile with hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy OR ≥ 12 months of amenorrhea and at least 50 years of age) are eligible to participate without the above precautions.
* Willing and able to comply with study procedures and requirements and attend all study visits as defined in this protocol.

Exclusion Criteria

Subjects with any of the following exclusion criteria will not be eligible for enrollment:

General Exclusion Criteria:

* Unable or unwilling to give informed consent.
* Pregnant or breast feeding
* Previous carpal tunnel release on the study hand
* History of steroid injection into carpal tunnel or surgery on the affected wrist within the past 6 months.
* Prisoners, institutionalized individuals, or others who may be considered vulnerable populations, such as individuals with dementia.

Laboratory Exclusion Criteria:

The following laboratory tests as indicated or as per clinical judgement:

* Bilirubin > 2.0; serum aspartate transaminase (AST) > 4 X upper limit of normal, or alanine aminotransferase (ALT) > 4 X upper limit of normal as a marker of liver disease
* Hemoglobin < 7g/dL; white blood cell count ≤2,000/mm3 (≤2.0 x 109/L) or ≥20,000/mm3 (≥20 x 109/L); platelet count ≤40,000/μL (≤40 x 109/L); absolute neutrophil count ≤1 x 109/L; lymphocyte count <0.3 x 109/L at screening as a marker of poor nutrition
* Plasma and/or serum fasting glucose > 300 or HbA1c > 9 as a marker of poor diabetic control
* Creatinine >2.5, cystatin c >3 or eGFR< 25 ml/min/1.73 m2 as a marker of advanced kidney disease,
* CRP > 10 or ESR >25 as a marker of systemic inflammation
* Unstable (as per clinical judgement) major cardiovascular, renal, endocrine, immunological, or hepatic disorder

Clinical History Exclusion Criteria

* History of diverticulitis or diverticulosis with GI bleeding, as per clinical judgement
* Any of the following clinical diagnosis or conditions: cervical radiculopathy, renal failure (see laboratory exclusion criteria), liver disease (see laboratory exclusion criteria), peripheral nerve disease, uncontrolled diabetes (see laboratory exclusion criteria), or other metabolic disorder; as per clinical judgement
* Human immunodeficiency virus infection
* Known active hepatitis B or C infection
* Invasive fungal infection
* Uncontrolled (as per clinical judgement) pleural/pericardial effusions or ascites
* New/active invasive cancer except non-melanoma skin cancers

Medication Exclusion Criteria

* Known hypersensitivity or allergy to Fisetin or other flavonoids
* Currently participating in another study using Fisetin or currently taking any flavonoid as a nutritional supplement. Note that consuming foods rich in flavonoids is NOT an exclusion, both because flavonoids are present in almost all fruits and vegetables, making such an exclusion impossible as a practical matter, and, from a scientific perspective, the amount of flavonoids in general, and Fisetin in particular, present in foods is far lower than the dose that will be administered in the trial.
* Patients currently taking medications listed in the Investigator Brochure are excluded unless medication can be safely held following the guidelines in the Investigator Brochure.
* If the patient is required to initiate any medication listed in the Investigator Brochure during the study, the PI will reassess their continued participation in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Amadio, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carpal Tunnel Syndrome: Adult men and women who had a clinical diagnosis for Carpal Tunnel Syndrome (CTS) received Fisetin for 2-day periods for 2 months.
  Fisetin: 100 mg capsules orally for 2 consecutive days and, after 1 month, another 2 consecutive days
Period: Overall Study
Arm/Group | Carpal Tunnel Syndrome
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carpal Tunnel Syndrome
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Boston Carpal Tunnel Syndrome (BCTQ) Score
Description: The Boston Carpal Tunnel Syndrome questionnaire (BCTQ) assesses symptom severity and overall function of subjects with Carpel Tunnel Syndrome. The questionnaire consists of two sections: 1. Symptom Severity (11 questions) and 2. Functional Status (8 questions). Subjects are asked to rate each question on a scale of 1 to 5. The mean score for each section is calculated by summing the individual question responses and diving by the number of questions resulting in a total score ranging from 1 to 5, with higher scores indicating greater symptom severity and dysfunction.
Time Frame: Baseline, 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carpal Tunnel Syndrome
Number analyzed (Participants) | 40
score on a scale | -0.5 (0.6)

2. Secondary Outcome: Percent Decrease in Blood Markers of Cellular Senescence, e.g., p16, IL-6, IL-15, TNF, PAI-1, ICAM-1, and Additional Exploratory, Novel Assays
Description: Blood samples collected to measure percent decrease in circulating blood biomarkers of senescence
Time Frame: Baseline, 60 days
Reporting Status: Not Posted

3. Secondary Outcome: Percent Decrease in Blood Markers of Cellular Senescence in Long-term
Description: percent decrease in blood markers of cellular senescence, e.g., p16, IL-6, IL-15, TNF, PAI-1, ICAM-1, and additional exploratory, novel assays
Time Frame: Baseline, 180 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of investigational product administration through post-treatment follow up, approximately 180 days.
Description: Adverse event definition used in this study: An untoward or undesirable experience associated with the use of a medical product (i.e., drug, device, biologic) in a patient or research subject.
  Adverse events were collected through specific questioning and/or examination.
Arm/Group | Carpal Tunnel Syndrome
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 15/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carpal Tunnel Syndrome (N=40)
Weight Gain (Investigations) | 1
Loose Bowels (Gastrointestinal disorders) | 1
Increased Pain (General disorders) | 7
Surgery due to Continued Pain (General disorders) | 6
C-Reactive Protein Level Increased (Investigations) | 1
Increased Symptom Severity (General disorders) | 5
Leg Cramping (Musculoskeletal and connective tissue disorders) | 1
Headaches (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05416515/Prot_SAP_000.pdf